CLINICAL TRIAL: NCT00078104
Title: Proinflammatory Gene Expression and Prostanoid Levels in a Clinical Model of Tissue Injury
Brief Title: Prostanoid Levels After Medication to Prevent Pain Following Third Molar (Wisdom Tooth) Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040124; 04-D-0124
Record Dates: First submitted 2004-02-18; First posted 2004-02-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Healthy; Tooth Extraction
Keywords: Prostanoid; Cyclooxygenase (COX); Selective Cox Inhibitor; Acute Peripheral Inflammation; Neuronal Expression of COX; Pain; Coxibs; Wisdom Teeth; Third Molar Extraction; Third Molar Impaction
MeSH Terms: conditions — Pain

INTERVENTIONS:
Procedure: Extraction of wisdom teeth

SUMMARY:
This study will evaluate how well different medications work to relieve pain following third molar (wisdom tooth) extraction. Scientists believe that hormone-like substances called prostanoids contribute to pain following oral surgery. Prostanoids are produced by cyclooxygenase (COX) enzymes. This study will examine how different medicines inhibit the COX enzymes and reduce the amount of prostanoids, and thus the amount of inflammation and pain. The study will also look at genetic factors involved in the production of prostanoids and the response to pain medication. (Only the bottom two wisdom teeth are extracted for this study. Patients whose top wisdom teeth also need to be removed will have those teeth extracted, also free of charge, at least 2 weeks after the first surgery.)

Healthy normal volunteers between 16 and 35 years of age who are in general good health and who require third molar extraction may be eligible for this study. Candidates are screened with a medical history and oral examination, including dental x-rays as needed to confirm the need for third molar removal.

On the morning of surgery, patients have blood drawn to obtain DNA for genetic study. Women of childbearing age have a urine pregnancy test. One hour before surgery, patients receive a dose of rofecoxib (Vioxx® (Registered Trademark)), acetaminophen (Tylenol® (Registered Trademark)), or placebo (a pill with no active ingredient). A half-hour before surgery, they receive either a standard painkiller called keterolac (Toradol® (Registered Trademark))) or placebo through an arm vein. All patients also receive the sedative midazolam (Versed® (Registered Trademark)), also through an arm vein, to induce drowsiness and a local anesthetic (lidocaine) to numb the mouth. After the mouth is numbed, but before the wisdom teeth are extracted, a biopsy (removal of a small piece of tissue) is conducted in the area of the cheek next to the wisdom tooth.

After the surgery, a small piece of tubing is placed into both extraction sites. Every 20 minutes for the next 3 hours, inflammatory fluid is collected from the tubing to measure chemicals that are believed to cause pain and swelling. Patients complete questionnaires every 20 minutes to rate their pain. Those who still have pain an hour after surgery may request and receive a "rescue drug" called tramadol (Ultram® (Registered Trademark)) for pain relief. Patients remain in the clinic from 3 to 6 hours to monitor the effects of the study drugs as the anesthetic wears off.

After surgery a second biopsy is done to measure any changes in the chemicals being produced in response to the surgery. For this biopsy, patients are assigned to one of two groups - one group has the second biopsy within 3 hours of surgery, before taking the rescue drug, and the other group returns to the clinic the next morning for a biopsy 24 hours after surgery. Patients in the second group leave the clinic after surgery with two pain medications (tramadol and the study drug) and forms to record pain ratings at home. They are permitted to take only the pain medications provided and only at certain times.

At the end of their participation in the study, all patients are given the pain medication flurbiprofen (Ocufen® (Registered Trademark)) to take at home.

DETAILED DESCRIPTION:
Two cyclooxygenase isozymes, COX-1 and -2, are known to catalyze the rate-limiting step of prostaglandin synthesis and are the targets of nonsteroidal anti-inflammatory drugs. Recently, the presence of a variant of COX-1, named COX-3, has been demonstrated that is especially sensitive to acetaminophen and strongly expressed in brain tissue. The proposed study will examine prostanoid suppression in the periphery by inhibition of COX-1, -2, and -3, and evaluate the time course of expression of COX isoenzymes in terms of level of mRNA and protein itself.

Subjects (N equals 88) will be healthy volunteers scheduled for the surgical removal of impacted third molars. Using a double-blinded, randomized, parallel study design, subjects will be allocated to one of four treatment groups and will be administered a dose of blinded medication or placebo. One hour prior to oral surgery, rofecoxib 50 mg, acetaminophen 1000 mg or placebo in two groups will be administered orally. Half hour prior to surgery, ketorolac 30 mg or placebo, will be administered intravenously. Microdialysis will be performed with sample collection concurrent with pain report over the immediate postoperative period of three hours, and the collected transudate will be analyzed by ELISA to evaluate prostanoid (prostaglandin E2, thromboxane B2) production. Subjects within each group will be further randomized to have a biopsy collected at baseline prior to surgery and either at the time when a subject asks for rescue drug within 3 hours or at 24 hours following surgery. The biopsies will be frozen in liquid nitrogen and assayed later by RT-PCR for levels of COX-1, COX-2, or COX-3 mRNA, and by microarray for evaluation of change in overall mRNA expression. A portion of the biopsy samples will be immunostained to reveal the tissue-specific pattern of each COX isoenzymes expression within the inflammatory tissue, and another part of the biopsy samples will be analyzed by Western blot to quantify the amount of protein. Fifty ml of blood will be collected from all subjects, and the single nucleotide polymorphisms (SNPs) in the genes regulated by inflammatory responses such as COX-1, COX-2, PGE receptors (EPs), and microsomal PGE synthase (mPGES) genes, will be analyzed to investigate the role of genetic factors in individual differences of drug responses. The analgesic effect of the drugs will be assessed in the clinic every 20 minutes for the first three hours after extractions, and on the next morning before taking any medication using two pain intensity assessment instruments: a category scale, and a visual analog scale (VAS).

We anticipate that non-selective COX inhibitor, the selective COX-2 inhibitor, and the selective COX-3 inhibitor will differentially alter prostanoid production over the time course evaluated, and that primary sensory neurons innervating in the inflammatory tissues may differentially express COX isoenzymes that differ in sensitivity to prototypic NSAIDs, coxibs, and acetaminophen. We also anticipate that several SNPs will contribute to the individual differences in COX expression and drug responses, which has implications for individual variation in pain, analgesic responses, and neuronal plasticity.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female volunteers referred for third molar extraction willing to undergo 2 or 3 visits: 1 screening visit; 1 surgical appointment; and possible 1 follow-up research-related appointment

Between the ages of 16 to 35 years (based upon eruption patterns and age-related complications associated with surgical extraction of third molars)

In general good health- American Society of Anesthesiologists (ASA) status I or II (healthy subjects based upon criteria for safe administration of out-patient conscious sedation)

Willing to undergo observation period for three hours postoperatively

Ability to complete a 100 mm visual analog scale and a category scale every 20 minutes for the first 3 postoperative hours

Willing to have a microdialysis probe placed beneath the surgical flap during the first 3 hours post-surgery

Willing to have a preoperative biopsy on the day of surgery, and a postoperative biopsy either within 3 hours or at 24 hours following surgery

Willing to return, if needed, 24 hours post-operation for the postoperative biopsy

Must have two lower partial bony impacted wisdom teeth fully covered by intact soft tissue (rating equals 3) or fully bony impacted (rating equals 4) wisdom teeth (mandibular third molars)

As assessed at the screening visit, the sum of the mandibular third molar surgical difficulty ratings must be between 6 to 8 in order to evaluate subjects experiencing similar pain levels

EXCLUSION CRITERIA:

Patients who are allergic to aspirin, NSAIDs, sulfites, or amide anesthetics

Patients who have had asthma, or hives

Patients who are pregnant or nursing

Patients with history of peptic ulcers and/or GI bleeding

Chronic use of medications confounding the assessment of the inflammatory response or analgesia, for example, NSAIDs, COX-2 inhibitors, antihistamines, steroids, antidepressants

Patients who have significant psychiatric history

Patients who have a clinical signs suggestive of infection, inflammation, or pre-existing pain at either extraction site

Patients with severe kidney disease

Patients who are taking any of the following drugs: ACE inhibitor; potassium sparing diuretics; aspirin on a near daily basis; coumadin or other blood thinners

Patients who are taking drugs known to inhibit P450 2C9 and drugs metabolized by P450 2D6

Patients who have G6PD deficiency and those taking St. John's Wort

Unusual surgical difficulty (determined from panoramic radiograph or during the actual surgery)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148
Dates: Start 2004-02; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bazan NG. COX-2 as a multifunctional neuronal modulator. Nat Med. 2001 Apr;7(4):414-5. doi: 10.1038/86477. No abstract available. PMID 11283664
- [Background] Butte A. The use and analysis of microarray data. Nat Rev Drug Discov. 2002 Dec;1(12):951-60. doi: 10.1038/nrd961. PMID 12461517
- [Background] Chandrasekharan NV, Dai H, Roos KL, Evanson NK, Tomsik J, Elton TS, Simmons DL. COX-3, a cyclooxygenase-1 variant inhibited by acetaminophen and other analgesic/antipyretic drugs: cloning, structure, and expression. Proc Natl Acad Sci U S A. 2002 Oct 15;99(21):13926-31. doi: 10.1073/pnas.162468699. Epub 2002 Sep 19. PMID 12242329